CLINICAL TRIAL: NCT00294021
Title: Long-term Impact of the Pneumococcal Conjugate Vaccine on Pneumococcal Nasopharyngeal Colonization and Immune Correlates for Disease Protection
Brief Title: Long-term Impact of Pneumococcal Conjugate Vaccine on Carriage
Status: Completed | Type: Observational
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Institute of Child Health (Other); Finnish Public Health Institute (Unknown); Thrasher Research Fund (Other); Grand Challenges in Global Health (Other)
Responsible Party: Principal Investigator, Katherine O'Brien, Professor, Johns Hopkins Bloomberg School of Public Health
Other Study IDs: CAIH-LTNP
Record Dates: First submitted 2006-02-17; First posted 2006-02-20 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2012-09

CONDITIONS: Pneumococcal Infections
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nasopharyngeal specimens will be collected for isolation of pneumococcus; saliva and serum specimens will be collected for antibody assays
Oversight: Data Monitoring Committee: No

SUMMARY:
Pneumococcus is a major cause of morbidity and mortality. In 2000, a pneumococcal conjugate vaccine (PCV) was licensed for use in children and is now part of the routine childhood vaccine schedule. PCV is known to reduce invasive disease and protect against nasopharyngeal (NP) acquisition of vaccine serotype pneumococci; it also results in an increased risk of nonvaccine serotype carriage. This study proposes to assess the longterm impact of vaccine on NP carriage in a setting where there is intense antibody pressure on the ecology of the pneumococcus. A cross sectional study of pneumococcal NP colonization among American Indian children will be combined with surveillance for invasive disease in the same population. The purpose is to determine the impact of community wide PCV use on NP colonization and the relationship with invasive disease. This longterm safety issue needs to be assessed to fully evaluate the impact of vaccine on NP ecology and invasive disease.

DETAILED DESCRIPTION:
There are four specific aims for this study: (1) to determine the overall and serotype specific prevalence and incidence of pneumococcal carriage among children and adults at high risk for carriage and disease in the era of routine pneumococcal conjugate vaccine (PCV) use compared with those measures in the same population prior to use of PCV vaccine; (2) to characterize the intrafamilial NP transmission of clones among those living with children less than 8 years of age; (3) to determine the immune correlates of protection from serotype specific pneumococcal carriage among individuals immunized and not immunized with PCV; and (4) to determine the relative invasiveness of serotypes of pneumococcus during an era of widespread PCV use and compare this to the relative invasiveness of serotypes prior to routine use of PCV.

ELIGIBILITY:
Inclusion Criteria for the Family to Participate.

1. At least one parent is a member of the Navajo or White Mountain Apache Tribe
2. Family home is on or near the Navajo or Apache reservation
3. At least one child in the household is 8 years of age or younger (minimum age of eligibility: birth)
4. At least one child in the household is fully immunized with Prevnar.
5. At least two people in the household will participate in the study
6. Willingness to participate for a 6-month time period

Exclusion Criteria for the Family to Participate.

1. Family will be moving off reservation during the study period

Inclusion Criteria for Individuals.

1. Living in the household
2. Willing to participate for a 6-month time period

Exclusion Criteria for Individuals.

1. Congenital anomalies of the nasopharynx

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adults and children living on the Navajo or White Mountain Apache reservations
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2006-03; Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine L O'Brien, MD, MPH, Principal Investigator — Johns Hopkins Center for American Indian Health
Locations (1):
- Johns Hopkins Center for American Indian Health, Chinle, Fort Defiance, Whiteriver, AZ; Gallup, Shiprock, NM, Arizona, United States